CLINICAL TRIAL: NCT06441734
Title: Iron Status in Autism Spectrum Disorders in Children Attending Assiut Pediatric University Hospital
Brief Title: Iron Status in Autism Spectrum Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, esraa hefzy shaker mostafa, principle investigator, Assiut University
Other Study IDs: anemia in autism
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group
  Interventions: Diagnostic Test: cbc serum ferritin serum iron
- control group
  Interventions: Diagnostic Test: cbc serum ferritin serum iron

INTERVENTIONS:
Diagnostic Test: cbc serum ferritin serum iron — by using sample of blood to do cbc and serum ferritin and serum iron during 1year

SUMMARY:
to evaluate the prevalence of iron deficiency anemia in group with autism spectrum disorders in comparison to normal children group

ELIGIBILITY:
Inclusion Criteria:

* children who are diagnosed with autism spectrum disorder according to DSM -V
* not having infection inflammatory conditions chronic physical illness
* children who are not receiving iron supplementation

Exclusion Criteria:

* age below 2 years and above 12 years
* having an infection or inflammatory conditions chronic physical illness
* receiving iron supplementation

Ages: 2 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: children age from 2years to 12 years not having an infection or inflammatory conditions or physical illness
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-08-02 (Estimated); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
iron status in autism spectrum disorders | 1 year
  by cbc serum ferritin serum iron

CONTACTS AND LOCATIONS:
Overall Officials: khalaf abdelaal said, lecturer, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Beltagi M. Autism medical comorbidities. World J Clin Pediatr. 2021 May 9;10(3):15-28. doi: 10.5409/wjcp.v10.i3.15. eCollection 2021 May 9. PMID 33972922
- See also: Related Info — http://www.ncbi.nlm.nih.gov